CLINICAL TRIAL: NCT00214344
Title: Evaluating the Usefulness of Preparing Families For Withdrawal of Mechanical Ventilation From Their Family Member: A Pilot Study
Brief Title: Family Preparation Study For Withdrawal of Mechanical Ventilation From Their Family Member
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: M-2003-0040
Record Dates: First submitted 2005-09-15; First posted 2005-09-21 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2005-09

CONDITIONS: Mechanical Ventilation; Critically Ill
Keywords: dying
MeSH Terms: conditions — Critical Illness

INTERVENTIONS:
Behavioral: family preparation for withdrawing life support

SUMMARY:
Using the self-regulation theory, an intervention to prepare families for that experience was developed. This study will assess the impact of the intervention on a family's evaluation of their preparation and their short-term coping. The site used for this study will be the Trauma and Life Support Center (TLC), University of Wisconsin (UW) Hospital. After a decision has been made to withdraw life support, a member of the TLC staff will approach the next of kin of the patient to inform him/her about the study and inquire about his/her interest to participate. Using an experimental design, 10 family members will be assigned to the control group and 10 to the intervention group. Upon agreement, a research nurse will use a "coin toss method" for group assignment of the subjects until there are ten in each group. Experimental group subjects will receive the intervention after the family meeting. Demographics of the next of kin will be collected at this time. Patient information such as demographics, diagnosis, and time of withdrawal and death will be collected too. Two to four weeks after death, a telephone interview will be conducted with the next of kin using the "Evaluation of the Experience of Withdrawal" questionnaire and the Profile of Mood State - shortened version.

Potential benefits are that the families will be prepared for the experience of the dying patient, which will help them cope better during withdrawal and after their loss. There are no major risks to the subjects but there might be an increase in psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* Next of kin of a patient who will have withdrawal of life support
* Participant must be 18 years of age or older and read, write, and speak English

Exclusion Criteria:

* Family is unusually highly emotional
* Patient will be a living donor
* Patient is conscious

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-10; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Are the families who received education/counseling better prepared for the experience of the dying patient

SECONDARY OUTCOMES:
This is a feasibility Pilot Study

CONTACTS AND LOCATIONS:
Overall Officials: Karin T Kirchhoff, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States